CLINICAL TRIAL: NCT01080196
Title: Reducing Falls With RENEW in Older Adults Who Have Fallen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Paul LaStayo, Primary Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 26292; R01AG031255-01A1 (NIH)
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Muscle Atrophy; Physical Deconditioning
Keywords: Falling risk; muscle conditioning; muscle size; isometric strength; Incidence in falls
MeSH Terms: conditions — Muscular Atrophy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RENEW (Experimental): RENEW will occur on a recumbent ergometer that appears like a normal stepper ergometer. While resisting the foot pedal movement the participant experiences eccentric muscle contractions about the knee and hip while performing negative work. The progression of the 3 x/week (every other day), 12 week RENEW program will be determined as a function of the rating of perceived exertion (RPE) using a "target" workload on the monitor. RENEW will be increased very slowly over the first 3 weeks and, subsequently, to maintain an 11-13 perceived exertion. During the formal RENEW training regimen the participants become fully acclimated to the device (week 3-4) the total RENEW load will increase weekly with no increase in their RPE.
  Interventions: Behavioral: RENEW
- TRADITIONAL (No Intervention): The TRAD group will perform their lower extremity resistance exercise for 15 minutes per session with isotonic weight machines and cuff weights as part of their multicomponent exercise fall reduction program (MCERFP). The progression of the 3 x/week, 12 week TRAD program will be determined as a relative function of their 1 repetition maximum (1RM) weight that can be lifted in a safe and successful manner. The 1RM will be measured before the 12 week training program and every 2 weeks thereafter. A "target" resistance workload (i.e., weight level) commensurate with 60-70% of the 1RM of the knee and hip extensors will be calculated bi-monthly and 3 sets of 15 repetitions of 3-4 different knee and hip exercises will be used over a 15 minute time period.

INTERVENTIONS:
Behavioral: RENEW — RENEW will occur on a recumbent ergometer that appears like a normal stepper ergometer. While resisting the foot pedal movement the participant experiences eccentric muscle contractions about the knee and hip while performing negative work. The progression of the 3 x/week (every other day), 12 week RENEW program will be determined as a function of the rating of perceived exertion (RPE) using a "target" workload on the monitor. RENEW will be increased very slowly over the first 3 weeks and, subsequently, to maintain an 11-13 perceived exertion. During the formal RENEW training regimen the participants become fully acclimated to the device (week 3-4) the total RENEW load will increase weekly with no increase in their RPE.
  Arms: RENEW

SUMMARY:
This clinical trial will compare the effects of a high intensity Resistance Exercise via Negative Work (RENEW) vs. Traditional resistance exercise (TRAD) as part of a mult-component exercise and fall-reduction program on muscle conditioning; falling risks; as well as the fall incidence in older adults who have fallen. We anticipate that muscle conditioning will mediate the effect of RENEW on falling risks and fall incidence.

DETAILED DESCRIPTION:
Muscle atrophy and weakness accompanying aging contributes greatly to an increased risk and incidence of falling. Over one-third of individuals 65 years of age or older experience a fall [1,2]. In a 2006 review [3] of 16 controlled (prospective and retrospective) studies [4-8] major factors affecting risk were identified with the most influential risk factors being muscle weakness, and deficits in balance and gait. The rate of muscle de-conditioning is accelerated by inactivity, muscle disuse and co-morbid conditions [9-12]. Older individuals with deficits in muscle size, strength and power can become so mobility-limited that simply walking to the mailbox is at the upper limit of their physical capacity [9] Hence, improving the muscle conditioning of an elderly individual with high fall risk may decrease the risk and incidence of falls [13-18]. Muscle conditioning often requires considerable effort, yet many elderly individuals lack the energetic reserves required for high-intensity exercise. Consequently, both elderly women and men are caught in a "downward-spiral" as their muscle de-conditioning accelerates the myriad risks of falling and the incidence of life-threatening falls.

We have explored the safety and feasibility of a high-intensity Resistance Exercise via Negative, Eccentrically-induced Work (RENEW) in multiple groups of de-conditioned elderly males and females, many characterized as being at-risk for a fall due to their impaired muscle condition, balance, mobility and confidence. Compared to traditional resistance exercise (TRAD), RENEW is novel and advantageous in that RENEW: is a high-intensity exercise for muscle, yet requires little effort (resulting in high levels of adherence); induces unprecedented muscle conditioning (size, strength and power); and lowers falling risks (balance, mobility and confidence) [19-23]. This study is unique and timely because it is unknown if RENEW's amplified muscle conditioning translates to a decreased incidence of falls, particularly for those at the highest risk for an injurious fall, i.e. those who have fallen. Further, RENEW's long-term sustainability has not been explored.

This clinical trial will compare the effects of RENEW vs. TRAD as part of a multi-component exercise and fall-reduction program (MCEFRP) on muscle conditioning (muscle size, strength, power); falling risks (balance, mobility and confidence); as well as the fall incidence. We anticipate that muscle conditioning will mediate the effect of RENEW on falling risks and fall incidence. As well, the sustained benefit of RENEW will be explored.

Objective #1: Test whether RENEW's effect is different than TRAD's effect on muscle conditioning, i.e., muscle size, strength and power.

• H1a: RENEW will result in greater increases (relative to TRAD) in whole muscle volume, isometric strength and concentric power of the leg extensor muscles, specifically the quadriceps.

Objective #2: Test whether the effects of RENEW on falling risks is mediated by muscle conditioning.

* H2a: RENEW will decrease falling risks (impaired balance, mobility and confidence) more than TRAD.
* H2b: RENEW's effects on falling risks will be mediated by greater muscle conditioning.

Objective #3: Determine if RENEW lowers fall incidence more than TRAD.

• H3a: The RENEW intervention will result in a lower fall incidence (falls and near falls) than TRAD via the direct influence on muscle conditioning and via the indirect influence of decreasing falling risks.

ELIGIBILITY:
Inclusion Criteria:

* male or a female at least 65 years of age or older with 2 or more self-reported co-morbid conditions.
* experienced at least 1 fall (defined for this study as unintentionally coming to rest on the ground, floor, or other lower level) in the previous 12 months
* ambulatory, community dwelling with gait speed ranging from of 25m/min to 80m/min
* medically cleared by their physician to participate in a 60 minute (with rests) MCERFP
* capable of performing RENEW on the ergometer (see below)
* recall of all 3 items (or 1-2 items with a normal clock drawing test) on the Mini-Cog instrument for dementia

Exclusion Criteria:

* progressive diagnosed neurologic disease (e.g., Parkinson's, multiple sclerosis, Guillain-Barre, Alzheimers)
* any dystrophies or rheumatologic conditions that primarily affects muscle (muscular dystrophy, PMR)
* having already participated in a MCEFRP
* regular (3x/week) aerobic or resistance exercise performed over the past 12 months; "aerobic" defined as hiking, fast-walking, jogging, running swimming or cycling; "resistance" defined as weight training with bands, cable, free-weights or weight-machines
* Any of the following list of absolute contraindications for MRI:
* Cardiac Pacemakers (except in rare, controlled environments)
* Cochlear (inner ear) implants
* Swan-Ganz catheters with thermodilution tips
* Ferromagnetic or unidentifiable aneurysm clips of the brain
* Implanted neuro stimulators
* Metal or unidentifiable foreign bodies in the eyes
* Shrapnel near a vital organ
* Extreme claustrophobia

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-04; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul C Lastayo, PT, PhD, Principal Investigator — Department of Physical Therapy, University of Utah
Locations (1):
- Department of Physical Therapy, University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] LaStayo P, Marcus R, Dibble L, Wong B, Pepper G. Eccentric versus traditional resistance exercise for older adult fallers in the community: a randomized trial within a multi-component fall reduction program. BMC Geriatr. 2017 Jul 17;17(1):149. doi: 10.1186/s12877-017-0539-8. PMID 28716003

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RENEW | TRADITIONAL
Started | 68 | 66
Completed | 68 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- TRADITIONAL: The TRAD group will perform their lower extremity resistance exercise for 15 minutes per session with isotonic weight machines and cuff weights as part of their MCERFP. The progression of the 3 x/week, 12 week TRAD program will be determined as a relative function of their 1 repetition maximum (RM) weight that can be lifted in a safe and successful manner. The 1RM will be measured before the 12 week training program and every 2 weeks thereafter. A "target" resistance workload (i.e., weight level) commensurate with 60-70% of the 1RM of the knee and hip extensors will be calculated bi-monthly and 3 sets of 15 repetitions of 3-4 different knee and hip exercises will be used over a 15 minute time period.
- Total: Total of all reporting groups
Arm/Group | RENEW | TRADITIONAL | Total
Number analyzed (Participants) | 68 | 66 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.59 (7.39) | 75.59 (6.98) | 76.1 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 42 | 87
  Male | 23 | 24 | 47
Region of Enrollment [Number; unit: participants]
  United States | 68 | 66 | 134

OUTCOME MEASURES:

1. Primary Outcome: The Number of Days Survived Without a Fall Over the 1 Year Duration of the Study
Time Frame: 12 months
Measure: Mean (Standard Error); unit: Days survived without a fall.
Arm/Group | RENEW | TRADITIONAL
Number analyzed (Participants) | 68 | 66
Days survived without a fall. | 239 (18) | 249.67 (16.38)

2. Other Pre Specified Outcome: Thigh Lean Tissue Cross Sectional Area (CSA) (cm^2)
Description: Magnetic resonance imaging (MRI) was used for determination of the cross-sectional area (CSA) (cm^2) of lean muscle mass. Bilateral MRI scans of the thighs were obtained in a coronal plane and the midpoint of the thigh was determined and defined as halfway between the superior margin of the femoral head and the inferior margin of the femoral condyles. Axial imaging (5 mm thick slices at 1 cm intervals) of the legs was then performed over 1/2 the length of the femur, centered at the midpoint of the thigh. Five images from the middle 1/3 of each thigh were used to determine average CSA of lean tissue.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: cm^2
Groups:
- RENEW: Resistance Exercise via Negative Work (RENEW) will occur on a recumbent ergometer that appears like a normal stepper ergometer. While resisting the foot pedal movement the participant experiences eccentric muscle contractions about the knee and hip while performing negative work. The progression of the 3 x/week (every other day), 12 week RENEW program will be determined as a function of the rating of perceived exertion (RPE) using a "target" workload on the monitor. RENEW will be increased very slowly over the first 3 weeks and, subsequently, to maintain an 11-13 perceived exertion. During the formal RENEW training regimen the participants become fully acclimated to the device (week 3-4) the total RENEW load will increase weekly with no increase in their RPE.
- TRADITIONAL: The Traditional (TRAD) group will perform their lower extremity resistance exercise for 15 minutes per session with isotonic weight machines and cuff weights as part of their MCERFP. The progression of the 3 x/week, 12 week TRAD program will be determined as a relative function of their 1 repetition maximum (RM) weight that can be lifted in a safe and successful manner. The 1RM will be measured before the 12 week training program and every 2 weeks thereafter. A "target" resistance workload (i.e., weight level) commensurate with 60-70% of the 1RM of the knee and hip extensors will be calculated bi-monthly and 3 sets of 15 repetitions of 3-4 different knee and hip exercises will be used over a 15 minute time period.
Arm/Group | RENEW | TRADITIONAL
Number analyzed (Participants) | 68 | 66
cm^2 | 92.6 [88.25 to 96.95] | 92.18 [87.88 to 96.47]

3. Other Pre Specified Outcome: Leg Extension Power (W)
Description: Leg extension power in watts (W) of each leg individually was measured on a Nottingham power rig. After three warm-up trials at 50%, 75%, and 100% effort, six test trials and the average of the three highest trials per leg were recorded.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: watts
Arm/Group | RENEW | TRADITIONAL
Number analyzed (Participants) | 68 | 66
watts | 104.73 [99.42 to 129.55] | 122.74 [108.3 to 137.18]

4. Other Pre Specified Outcome: Activities Specific Balance Confidence (ABC) (%)
Description: Self-reported level of balance confidence was assessed with the Activities Specific Balance Confidence (ABC) Scale. This 16-item questionnaire asks participants to score their level of confidence in performing situation-specific activities such as "reaching at eye level," "reaching on tiptoes," "picking up slipper from floor," and "walking in crowded mall" "without losing . . . balance or becoming unsteady." Each item is scored from 0 to 100%, with 0% being no confidence and 100% being full confidence in the ability to perform the activity without losing balance. The total ABC Scale score is the average sum of the individual item scores.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: percent
Arm/Group | RENEW | TRADITIONAL
Number analyzed (Participants) | 68 | 66
percent | 82.25 [76.82 to 87.68] | 80.93 [75.73 to 86.13]

5. Other Pre Specified Outcome: Six Minute Walk (6 MW) Test
Description: The 6 min walk (6 MW) test, a measure of the distance (m) a subject walks in 6 min, was used to assess overall mobility. Self-selected gait-speed was measured over a 50-ft course. Individuals were instructed to walk at a comfortable pace starting at the word "go." They were asked to walk out 25-ft and back. Timing took place from the command "go" until the starting line was crossed on the way back. Participants were allowed to use any walking aid they used on a daily basis.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | RENEW | TRADITIONAL
Number analyzed (Participants) | 68 | 66
meters | 439.18 [394.65 to 487.72] | 438.15 [397.39 to 478.92]

ADVERSE EVENTS:
Arm/Group | RENEW | TRADITIONAL
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/66
Other Adverse Events (participants affected / at risk) | 4/68 | 3/66
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RENEW (N=68) | TRADITIONAL (N=66)
joint and muscle pain (Musculoskeletal and connective tissue disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No